CLINICAL TRIAL: NCT06148909
Title: A Pilot Study on Small Talk Intervention With MI in Assisting Smokers to Quit
Brief Title: Small Talk Intervention With MI for Smoking Cessation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Small talk_smoking cessation
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Smoking Cessation; Motivation
Keywords: Smoking Cessation; Motivational Interviewing; Small Talks
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small Talk Motivational Interviewing (STMI) (Experimental): during the 8 session of smoking cessation, the first three sessions will be used to do small talks with the participant. And then from the fourth session onwards, the RA will add 30 minutes of MI about smoking cessation after engaging in small talk.
  Interventions: Other: Small Talk Motivational Interviewing
- Control (only MI) (No Intervention): Another two RA with at least one-year experience on counselling will be delivering the control group. Participant will receive MI for 30 minutes in each of the first three sessions and 1 hour in each of the remaining sessions. The control group will also receive the same duration and content of boosters as in the intervention group.

INTERVENTIONS:
Other: Small Talk Motivational Interviewing — Combining small talks and skills on Motivational Interviewing in the smoking cessation services
  Arms: Small Talk Motivational Interviewing (STMI)

SUMMARY:
The goal of this pilot study is to examine the effectiveness of the STMI in promoting abstinence in unmotivated smokers. The main questions it aims to answer are:

* Do unmotivated smokers treated with STMI exhibit higher abstinence rate than those in the control group?
* Do unmotivated smokers treated with STMI show higher intention to quit than those in the control group?
* Do unmotivated smokers treated with STMI show higher smoking reduction rates than those in the control group?
* Do unmotivated smokers treated with STMI show lower level of depressive symptoms than those in the control group?
* Do unmotivated smokers treated with STMI show higher adherence than those in the control group?
* Does STMI show higher consent rates than those the control?
* How does STMI affect the smoking behaviors in unmotivated smokers?

Participants will be randomized to (1) STMI or (2) control group for smoking cessation services via telephone, and then be invited to join a semi-structured interview.

DETAILED DESCRIPTION:
Two RAs with at least 1 year of experience in counseling or related work will be hired to deliver the intervention. The same RA will deliver the eight-session intervention weekly via telephone to the same participant within 2 months. The intervention contains eight sessions which is similar to that in YQL. Interventions will be delivered via telephone because YQL also used the same delivery mode to successfully contact and assist a considerable number of smokers to quit . Based on our team's experience in YQL, each session will last from 30 minutes to 1 hour.

In the first to third sessions, the RA will engage in small talk with the participants for 30 minutes. The RA will talk to the participants on the proposed topics including the weather, activities the participant engaged in last week and at weekends, music, food, and other hobbies, all of which were recommended in previous literature as topics that interest most people and create curiosity and enjoyment rather than animosity. From the fourth session onwards, the RA will add 30 minutes of MI about smoking cessation after engaging in small talk. During MI delivery, the RA will use core MI skills, including open-ended questions, affirmation, reflective listening, and summary, elicit-provide-elicit, evoking change talk, and roll with resistance to move the participants from engaging (first process of MI) to planning (last process of MI), as in YQL and other smoking cessation projects that use MI. The RA will aim to go through the engaging process in the fourth session, focusing process in the fifth session, focusing and evoking in the sixth session, and evoking and planning in the seventh and eighth sessions. When transitioning from small talk to MI, some simple transitional sentences are suggested, such as: "We have been talking for quite a while since our contact at the first time. Actually, I am quite interested in understanding your smoking behaviors. Do you mind talking with me about that?" If the participants refuse, the RA will continue to deliver small talk and repeat asking in the next session if the participants can move to talk about smoking or not.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-25 years old
* Have smoked any smoking products in the past 30 days
* do not intend to quit in the coming 30 days
* did not have a past-year quit attempt lasting for 24 hours or more
* are not currently in any smoking cessation programs
* are able to speak Cantonese and read Chinese

Exclusion Criteria:

* self-report having identified cognitive problems or psychosis, including schizophrenia, psychotic depression, and schizoaffective disorder will be excluded

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
biochemically-validated abstinence rate | 6-month follow-up
  participants will be invited to join a breath test at 6-month time point after they joined the study, to determine if they have quitted smoking or not

SECONDARY OUTCOMES:
Self-reported questionnaire | 1-week, 1-, 3-, 6-, 9-, and 12-month follow-ups
  Including self-reported quit rate, intention to quit, smoking reduction, depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ka Wai Katherine Lam, Phd, Principal Investigator — the polytechnic university of hong kong
Locations (1):
- Katherine Lam, Hong Kong, Hong Kong,China, Hong Kong